CLINICAL TRIAL: NCT04621188
Title: A Phase II Single-group Assignment, Multicenter Study of Efficacy and Safety of Lorlatinib Monotherapy After Failure of First-line Tyrosine Kinase Inhibitor in Patients With Advanced ROS1-positive Non-small Cell Lung Cancer (ALBATROS)
Brief Title: Lorlatinib After Failure of First-line TKI in Patients With Advanced ROS1-positive NSCLC (ALBATROS)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-2003; 2024-512028-12-00 (EU CTIS Number)
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: IFCT; ALBATROS; NSCLC; ROS1-positive; monotherapy
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lorlatinib (Experimental): 100 mg once daily
  Interventions: Drug: Lorlatinib

INTERVENTIONS:
Drug: Lorlatinib — 100 mg once daily

SUMMARY:
ROS1 rearrangements are present in 1-2% of NSCLC cases and define a distinct molecular subgroup. Like ALK (anaplastic lymphoma kinase) rearrangements in NSCLC, ROS1 fusions confer sensitivity to the inhibitor crizotinib. Crizotinib, which is a tyrosine kinase inhibitor (TKI), has been shown to be effective in tumors in several retrospective studies.

Recently the FDA approved entrectinib for the treatment of patients with ROS1-positive metastatic NSCLC. This indication is based on the results of pooled data from several trials. Together, these studies demonstrate the efficacy for entrectinib across a variety of solid tumor types including NSCLC with ROS1 fusion.

However, despite the efficacy of crizotinib or entrectinib in ROS1-positive NSCLC, patients will develop resistance to these tyrosine kinase inhibitors.

Lorlatinib is a new and potent ROS1 / ALK inhibitor optimized to penetrate the blood-brain barrier. A recent study has investigated the activity of lorlatinib against the crizotinib-resistant ROS1G2032R mutation. In this situation, lorlatinib effectively inhibited the catalytic activity of recombinant ROS1G2032R resulting in an antiproliferative response. Because of its potency as an ROS1 inhibitor and its ability to suppress the resistant ROS1 mutations, lorlatinib could be a treatment of choice in ROS1-positive NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent: Subjects must have signed and dated an IRB/IEC approved written informed consent form in accordance with regulatory and institutional guidelines. This must be obtained before the performance of any protocol related procedures that are not part of normal subject care. Subjects must be willing and able to comply with scheduled visits, treatment schedule, and laboratory testing
* Patients with histologically or cytologically confirmed diagnosis of locally advanced not eligible to a local treatment or metastatic NSCLC (Stage IIIB, IIIC or IV accordingly to 8th classification TNM, UICC 2015) that carries an ROS1 rearrangement, as determined by the molecular biology platform of the investigator by FISH assay or by Immunohistochemistry (IHC), or Next Generation Sequencing (NGS) or RNA sequencing approach.
* Disease Status Requirements: Disease progression meeting RECISTv1.1 after one prior line of treatment with crizotinib or entrectinib (+ one line of chemotherapy with or without immunotherapy before TKI treatment).

Note: patient with disease progression after treatment with another ROS1-TKI may still be eligible upon discussion with IFCT.

* Tumor Requirements: All Patients must have at least one measurable target lesion according to RECIST v1.1. The radiological assessment has to be done within the timelines indicated. In addition, patients with asymptomatic and neurologically stable CNS metastases (including patients controlled with stable or decreasing steroid use within the last week prior to study entry) will be eligible. The brain metastases may be newly diagnosed after disease progression with crizotinib or entrectinib or be present as progressive disease after surgery, whole brain radiotherapy or stereotactic radiosurgery (see Exclusion Criterion for the lapsed time period required between the end of radiotherapy and study entry). Patients who have leptomeningeal disease (LM) or carcinomatous meningitis (CM) will be eligible if the LM/CM is visualized on MRI or if documented baseline cerebral spinal fluid (CSF) positive cytology is available and asymptomatic and neurologically stable (including patients controlled with stable or decreasing steroid use within the last week prior to study entry).
* Tumor Sample Requirement: Tumour biopsy sampling on fresh tissue (FFPE blocks required) obtained after progression on crizotinib or entrectinib. Tumour biopsy should be exploitable for molecular analysis. If the tumour biopsy is not exploitable, the inclusion will be allowed if two blood samples are provided for tumoral cfDNA analysis. The Sponsor will monitor a posteriori the exploitability of provided tumour biopsies and will investigate the impossibility to perform or repeat tissue tumor sampling.
* Age ≥18 years.
* Life expectancy of at least 12 weeks, in the opinion of the Investigator.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) ≤ 2
* Adequate Bone Marrow Function, including: Absolute Neutrophil Count (ANC) ≥1.5 x 109/L; Platelets ≥100 x 109/L; Hemoglobin ≥9 g/dL.
* Adequate Pancreatic Function, including: Serum lipase ≤1.5 x ULN.
* Adequate Renal Function, including: Serum creatinine ≤1.5 x ULN or estimated creatinine clearance ≥45 mL/min as calculated using the method standard for the institution.
* Adequate Liver Function, including: Total serum bilirubin ≤1.5 x ULN; Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) ≤2.5 x ULN; ≤5.0 x ULN if there is liver metastases involvement.
* Participants must have recovered from treatment toxicities to CTCAE Grade ≤ 1 (for participants who have developed interstitial lung disease [ILD], they must have fully recovered) except for AEs that in the investigator' judgment do not constitute a safety risk for the patient.
* Participants must have recovered from effects of any major surgery, or significant traumatic injury, at least 35 days before the first dose of lorlatinib
* For all females of childbearing potential, a negative pregnancy test must be obtained within the screening period. A patient is of childbearing potential if, in the opinion of the investigator, she is biologically capable of having children and is sexually active. Additionally, all females of childbearing potential must provide an agreement to remain abstinent or use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for at least 90 days after the last dose of study drug.
* For men: agreement to remain abstinent or use an effective method of contraception (e.g., condom) during the treatment period and for at least 14 weeks after the last dose of study drug and agreement to refrain from donating sperm during this same period.
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study.
* Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedure.
* Participant has national health insurance coverage.
* Washout period: if previous progression on ROS1-TKI: 7 days from last dose of the drug. The washout period may be shortened to 2 days at investigator discretion.

Exclusion Criteria:

* Participants with disease progression on front-line treatment with TKI i.e. crizotinib or entrectinib limited to CNS or one non-CNS site (oligo-metastasis) and eligible to a local ablative treatment (surgery or stereotaxic radiotherapy).
* Histological transformation with neuro-endocrine differentiation.
* Spinal cord compression is excluded unless the patient demonstrates good pain control attained through therapy and there is stabilization or recovery of neurological function for the 4 weeks prior to study entry.
* Patients with symptomatic and neurologically instable CNS metastases or leptomeningeal metastasis (including patients that require increasing doses of steroids within one week prior to Day 0 of screening phase and during the screening phase to manage CNS symptoms).
* Major surgery within 35 days of study entry. Minor surgical procedures (eg, port insertion, mediastinoscopy, surgical procedure for re-sampling) are not excluded, but sufficient time at investigator discretion should have passed for wound healing.
* Radiation therapy within 2 weeks of study entry (except palliative to relieve bone pain). Palliative radiation (≤15 fractions) must have been completed at least 48 hours prior to study entry. Stereotactic or small field brain irradiation must have completed at least 2 weeks prior to study entry. Whole brain radiation must have completed at least 4 weeks prior to study entry.
* Prior therapy with an antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways, including, but not limited to, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4.
* Active and clinically significant bacterial, fungal, or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness.
* Clinically significant cardiovascular disease (that is, active or <3 months prior to enrollment): cerebral vascular accident/stroke, myocardial infarction, unstable angina, congestive heart failure (New York Heart Association Classification Class ≥ II), second-degree or third-degree AV block (unless paced) or any AV block with PR >220 msec.
* Ongoing cardiac dysrhythmias of NCI CTCAE Grade ≥2, uncontrolled atrial fibrillation of any grade, bradycardia defined as <50 bpm (unless patient is otherwise healthy such as long-distance runners, athletic patients etc.), machine-read ECG with QTc >470 msec, or congenital long QT syndrome.
* Patients with predisposing characteristics for acute pancreatitis according to investigator judgment (eg, uncontrolled hyperglycemia, current gallstone disease, alcoholism [more than 4 drinks on any day or 14 drinks per week where 1 drink is defined as the alcoholic beverage containing approximately 14 grams of pure alcohol, eg, 12 fl oz/360 mL regular beer or 5 fl oz/150 mL of wine] in the last month.
* History of bilateral or Grade 3 or 4 interstitial fibrosis or diffuse interstitial lung disease. Patients with history of prior radiation pneumonitis are not excluded.
* Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Evidence of active malignancy (other than current NSCLC, non-melanoma skin cancer, in situ cervical cancer, papillary thyroid cancer, DCIS of the breast or localized and presumed cured prostate cancer) within the last 3 years.
* Active inflammatory gastrointestinal disease, chronic diarrhea, symptomatic diverticular disease or previous gastric resection or lap band.
* Current use or anticipated need for food or drugs prohibited (see chapter 7.9 for details).
* Patients presenting with abnormal Left Ventricular Ejection Fraction (LVEF) by echocardiogram or Multi-Gated Acquisition Scan (MUGA) according to institutional lower limits.
* Breastfeeding female patients (including patients who intend to interrupt breastfeeding).
* Liver disease characterized by: ALT or AST level > 3 the upper normal limit (UNL) (≥ 5 x UNL for patients with liver metastases) confirmed on 2 consecutive measures OR impaired excretory function (e.g.. hyperbilirubinemia) or synthetic function or other conditions of decompensated liver disease e.g.: coagulopathy, Hepatic encephalopathy, hypoalbuminemia, ascites and bleeding from esophageal varices OR Acute viral or autoimmune or other types of hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) at 8 weeks by investigators | 8 weeks
  ORR is defined as the percentage of subjects with a confirmed complete response (CR) or partial response (PR) as per RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) at 8 weeks by Independent Reviewer Committee (IRC) | 8 weeks
  Percentage of subjects with a confirmed at 16 weeks complete response (CR) or partial response (PR) as per RECIST v1.1 criteria.
Progression Free Survival (PFS) | Up to 24 months
  Time between the date of first dose of study drug and the first date of documented disease progression (according to RECIST v1.1) or death (from any cause)
Time to progression (TTP) | Up to 24 months
  Time from the date of first dose of study drug to the earliest date of disease progression (according to RECIST v1.1.)
Disease control rate (DCR) at 8 weeks weeks) | 8 weeks
  Proportion of patients have achieved a confirmed best overall response of CR, PR or SD (Stable Disease) (according to RECIST v1.1.)
Duration of response (DOR) first documented response (CR or PR) to the earliest date of disease progression, or death due to any cause. | Up to 24 months
  Time from the date of the first documented response (CR or PR) to the earliest date of disease progression or death due to any cause.
Overall survival (OS) months | 12 months and 24 months
  Time from the date of first dose of study drug to the date of death due to any cause
Central Nervous System (CNS) Objective response rate (C-ORR) | Up to 24 months
  ORR estimated in patients with measurable CNS metastases at baseline.
CNS duration of response (C-DOR) measurable CNS metastases at baseline. | Up to 24 months
  DOR estimated in patients with measurable CNS metastases at baseline.
Time to CNS progression | Up to 24 months
  In patients without brain metastases baseline.
Change from baseline of EuroQol Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L) | Up to 24 months
  At all scheduled time points

CONTACTS AND LOCATIONS:
Overall Officials: Denis Moro-Sibilot, Study Chair — Grenoble - CHU; Michael Duruisseaux, Study Chair — Lyon - URCOT
Locations (34):
- France (34):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Centre Paul Papin, Angers
  - Angers - CHU, Angers
  - Annecy - CH, Annecy
  - Antony - Hôpital privé, Antony
  - Avignon - CH, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Bordeaux - CHU, Bordeaux
  - Bordeaux - Institut Bergonie, Bordeaux
  - Bordeaux - Polyclinique, Bordeaux
  - AP-HP Hôpital Ambroise Paré, Boulogne
  - Caen - CHU Côte de Nacre, Caen
  - Chauny - CH, Chauny
  - Cholet - CH, Cholet
  - Clermont-Ferrand - CHU, Clermont-Ferrand
  - Colmar - CH, Colmar
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Dijon - CRLCC, Dijon
  - CHRU Grenoble, Grenoble
  - Centre Hospitalier - Pneumologie, Le Mans
  - Hôpital Calmette, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - GRH Mulhouse Sud-Alsace, Mulhouse
  - AP-HP Hôpital Cochin, Paris
  - AP-HP Hopital Tenon - Pneumologie, Paris
  - Lyon - URCOT, Pierre-Bénite
  - Rouen - CHU, Rouen
  - Nouvel Hôpital Civil - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Hôpital Foch, Suresnes
  - CHU Toulouse - Pneumologie, Toulouse
  - CHU Bretonneau, Tours
  - Valenciennes - Clinique, Valenciennes
  - Vandoeuvre-lès-Nancy - CHU, Vandœuvre-lès-Nancy

REFERENCES:
- See also: Description IFCT website — http://www.ifct.fr/index.php/fr/la-recherche/item/2215-ifct-2003-albatros